CLINICAL TRIAL: NCT02130076
Title: The Effect of Interruption of TNFi on Endothelial Function in Patients With Rheumatoid Arthritis
Brief Title: Interruption of TNFinhibitors and Endothelial Function
Acronym: POET-VEF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, G. Rongen, Prof dr G Rongen, Radboud University Medical Center
Other Study IDs: IMM11-0103
Record Dates: First submitted 2013-01-08; First posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Reumatoid Arthritis; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Stop: Patients with stable RA stopping TNF inhibition
- Continue: Patients with stable RA continuing TNFi therapy

SUMMARY:
Patients with rheumatoid arthritis (RA) have an increased risk of cardiovascular events. This increased risk is thought to be driven by inflammation-induced endothelial dysfunction, an initial step in atherogenesis. Treatment with TNFalpha inhibitors (TNFi) improve endothelial function in patients with RA. Discontinuation of TNFi could therefore worsen endothelial function even in the absence of recurrence of systemic inflammation or reactivation of arthritis. If stopping TNFi results in worsening of endothelial function this would strongly suggest a higher cardiovascular risk in association with TNFi-wthdrawal

DETAILED DESCRIPTION:
Patients with rheumatoid arthritis (RA) have an increased risk of cardiovascular events. This increased risk is thought to be driven by inflammation-induced endothelial dysfunction, an initial step in atherogenesis. Both systemic as well as local (intra-arterial) treatment with anti-TNF-antibody therapy improves endothelial function in patients with vasculitis or RA as reflected by the vasodilator response to intra-arterially infused acetylcholine. Also other vascular functions that are (at least partially) endothelium-dependent such as flow-mediated dilation of the brachial artery and pulse wave velocity are improved when active RA patients are being treated with methotrexate plus TNFi, i.e. infliximab or etanercept. ( Therefore one may hypothesize that when TNFi therapy is stopped, endothelial function may worsen even in the absence of recurrence of systemic inflammation or reactivation of arthritis. Endothelial function tests are a marker of long-term cardiovascular mortality. If stopping TNFi results in worsening of endothelial function this would strongly suggest a higher cardiovascular risk in association with TNFi-wthdrawal. These findings would indicate an important drawback for stopping TNFi in RA patients.

To date it is unclear whether the worsening of endothelial function occurs within half a year following the (successful) cessation of TNFi, whether this decline occurs simultaneously, or prior to RA exacerbation and whether this deterioration process is delayed by additional use of statin and/or ACEi.

To improve cardiovascular prognosis in RA significantly it is important to increase our knowledge regarding these processes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent for POEET trial and this additional study
* On stable medication (except for TNFi-therapy)

Exclusion Criteria:

* Uncontrolled hypertension (RR > 140/90 mmHg average of three measurements at screening after 5 minutes of supine rest)
* Diabetes mellitus
* Heart failure or any other cardiovascular disease that is expected to induce changes in cardiovascular medication during the study period.
* Expected to start or change medication that can alter endothelial function (lipid lowering drugs, blood pressure lowering drugs, NSAIDs, immunosuppressive therapy other than TNFi drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable rheumatoid arthritis who are included in another study (POEET) to stop or continue their TNFi therapy.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Response to acetylcholine | 6 months
  The primary endpoint is the interaction between TNFi-withdrawal and the vasodilator response to acetylcholine expressed as difference in FBF between the withdrawal group and the continuing group.

SECONDARY OUTCOMES:
TNFi withdrawal and response to nitroprusside | 6 months
  Secondary endpoints are the interaction between TNFi-withdrawal and the vasodilator response to nitroprusside (expressed as difference in FBF between the withdrawal group and the continuing group). The response to SNP serves as an internal vasodilator control to assess potential endothelium-independent effects of TNFi-withdrawal on the response to acetylcholine.
VCAM and SCAM | 6 months

REFERENCES:
- [Derived] Rongen GA, van Ingen I, Kok M, Vonkeman H, Janssen M, Jansen TL. Vasodilator function worsens after cessation of tumour necrosis factor inhibitor therapy in patients with rheumatoid arthritis only if a flare occurs. Clin Rheumatol. 2018 Apr;37(4):909-916. doi: 10.1007/s10067-017-3961-6. Epub 2018 Jan 7. PMID 29307093